CLINICAL TRIAL: NCT05890508
Title: Electro-acupuncture for Long Covid Neuropsychiatric Symptoms: a Prospective, Randomized Sham-controlled, Double-blinded Clinical Trial
Brief Title: Electro-acupuncture for Long Covid Neuropsychiatric Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Zhong Lidan, Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021HMRF
Record Dates: First submitted 2023-06-01; First posted 2023-06-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Long Covid19; Neuropsychiatric Symptoms; Electro-acupuncture
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All patients and the investigators including the research assessors, the statistician, and the researchers interacting with the patients except the one who conducts the acupuncture therapy will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-acupuncture group (Experimental): The electro-acupuncture intervention will be conducted for 2 session per week during 16-week treatment duration, and will be followed up for 8 weeks. In this study, 7 acupoints are chosen:GV20(Baihui), EX-HN1(Sishencong), EX-HN3(Yintang), SP6(Sanyinjiao), ST36(Zusanli), ST40(Fenglong), and LR3(Taichong). The puncture is made in accordance with the standards of traditional Chinese medicine, to a depth of 1 to 3 cm depending on the thickness of the local tissues. The acupoints are subjected to 2-5 Hz electroacupuncture from an electroacupuncture device at an intensity (5 to 10 mA) that can produce a muscle twitch acceptable to the participant.
  Interventions: Device: Acupuncture
- Sham-acupuncture group (Sham Comparator): For subjects assigned to the sham control group, Streitberger's non-invasive acupuncture needles (Gauge 8 x 1.2/ 0.30 x 30mm) will be applied to serve as a sham control at the corresponding non-acupoints, leave 0.5 cun from the corresponding acupoints, with the same stimulation modality. Addtionally, the stimulation will be a "pseudo stimulation", which will be given by connecting the needle to the incorrect output socket of the electrical acupuncture stimulation instrument. The credibility and validity of this system have been well demonstrated.
  .
  Interventions: Device: Sham-acupuncture

INTERVENTIONS:
Device: Acupuncture — Disposable acupuncture needles (0.20 mm in diameter) are are used in the study. The acupoints are GV20(Baihui), EX-HN1(Sishencong), EX-HN3(Yintang), SP6(Sanyinjiao), ST36(Zusanli), ST40(Fenglong), and LR3(Taichong). Electrical stimulation will be delivered with waves at 2-5 Hz from an electroacupuncture device. The needles will be retained in position for 30 minutes.
  Arms: Electro-acupuncture group
Device: Sham-acupuncture — Streitberger's non-invasive acupuncture needles (Gauge 8 x 1.2"/ 0.30 x 30mm) will be applied to serve as a sham control at the same acupoints with the same stimulation modality and then connecting the needle to the incorrect output socket of the electrical acupuncture stimulation instrument. The sham points are "pseudo stimulation".
  Arms: Sham-acupuncture group

SUMMARY:
In this study, a 16-week randomized, sham-controlled, double-blinded clinical trial will be conducted to to investigate the efficacy and safety of electro-acupuncture compared to sham acupuncture for treatment of long covid neuropsychiatric symptoms.

DETAILED DESCRIPTION:
This is a prospective, randomized, sham-controlled, double-blinded and multiple center trial on electro-acupuncture for treating neuropsychiatric symptoms in long covid patients. A total of 150 participants will be randomly assigned to the electro-acupuncture and the sham-control group with 1:1 ratio. Both groups will receive 32 sessions of interventions during 16-week treatment duration (2 session per week), and will be followed up for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years of age to 80;
* history of SARS-CoV-2 PCR+ at least 4 weeks prior to study entry; SARS-CoV-2 negative (PCR) at study entry;
* at least one persistent neurological symptom (impaired concentration, headache, sensory disturbances, or depression, or "brain fog") that began around the time of the acute COVID-19;
* willing and able to consent, complete all assessment and study procedures.

Exclusion Criteria:

* any chronic or remote neurological disorder (i.e. stroke, head trauma, epilepsy, tumor);
* intellectual disability pre-existing to the Covid-19 episode;cardiovascular diseases such as arrhythmia, heart failure, myocardial infarction, and patients with cardiac pacemakers,
* acute brain injury or acute encephalopathy from another aetiology than covid (e.g., sepsis, liver or renal failure, alcohol or drug withdrawal, drug toxicity);
* documented pre-existing history of psychiatric illness, including substance abuse;
* open-heart cardiac surgery or cardiac arrest during the last 6 months;
* current hospitalization;
* pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive score on the Chinese version of the Mini-Mental State Examination (MMSE) scale | At baseline (before intervention), at 4, 8, 12, 16 weeks (the end of intervention) and 2 months after intervention (the end of follow-up).
  The MMSE can evaluate of five different domains of cognitive functions: (1) Orientation, with a maximum of 10 points, (2) Memory, with a maximum of 6 points, (3) Attention and calculation, with a maximum of 5 points, (4) Language, with a maximum of 8 points, and (5) Design copying, with a maximum of 1 point. It has a maximum score of 30, with MMSE score denotes severity of cognitive impairment as follows; mild: MMSE 21 to 24, moderate: MMSE 10 to 20, severe: MMSE less than 10.
Depression on the Chinese Beck Depression Inventory (CBDI) | At baseline (before intervention), at 4, 8, 12, 16 weeks (the end of intervention) and 2 months after intervention (the end of follow-up).
  The scale has a total of 21 questions, with an overall score of 63, 14-19 being mild depression, 20-28 being moderate depression, and above 29 being severe depression.

SECONDARY OUTCOMES:
Score of Insomnia Severity Index (ISI) | At baseline (before intervention), at 4, 8, 12, 16 weeks (the end of intervention) and 2 months after intervention (the end of follow-up).
  The Insomnia Severity Index in Chinese includes 5 questions to assess the severity and impact of insomnia, on an 0 to 4 scale, with the higher score reflecting worse insomnia symptoms.
Score of Brief Fatigue Inventory-Taiwanese (BFI-T) Form | At baseline (before intervention), at 4, 8, 12, 16 weeks (the end of intervention) and 2 months after intervention (the end of follow-up).
  BFI-T form is to assess the severity of fatigue and the impact of fatigue on daily functioning. Scoring Respondents rate each item on a 0-10 numeric scale, with 0 meaning "no fatigue" and 10 meaning "fatigue as bad as you can imagine." Scores are categorized as Mild (1-3), Moderate (4-6), and Severe (7-10).
Score of the Short Form 12 (SF12) | At baseline (before intervention), at 4, 8, 12, 16 weeks (the end of intervention) and 2 months after intervention (the end of follow-up).
  The SF-12V2 is a widely used generic HRQoL instrument, and its Chinese version has been validated and normed in the general Chinese population in Hong Kong. It consists of 12 questions measuring eight domains of health, including physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The scores are generated using an algorithm to generate a combined physical and mental health score for comparison with normative data. In the normative data: 1) the mean score was set to 50; 2) a score > 50 indicated better physical or mental health than the mean; 3) a score < 50 indicated worse physical or mental health than the mean.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Jue Wei, MD, Study Chair — Hong Kong Baptist University
Locations (1):
- Zhong Lidan, Kowloon Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Johns Hopkins University of Medicine Coronavirus Resource Center . COVID-19 Dashboard by the Center for Systems Science and Engineering (CSSE) at Johns Hopkins University (JHU). 2022. https://coronavirus.jhu.edu/map.html(16 February 2022, date last accessed)
- [Background] Spudich S, Nath A. Nervous system consequences of COVID-19. Science. 2022 Jan 21;375(6578):267-269. doi: 10.1126/science.abm2052. Epub 2022 Jan 20. PMID 35050660
- [Background] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937
- [Background] Crook H, Raza S, Nowell J, Young M, Edison P. Long covid-mechanisms, risk factors, and management. BMJ. 2021 Jul 26;374:n1648. doi: 10.1136/bmj.n1648. PMID 34312178
- [Background] Evans RA, McAuley H, Harrison EM, Shikotra A, Singapuri A, Sereno M, Elneima O, Docherty AB, Lone NI, Leavy OC, Daines L, Baillie JK, Brown JS, Chalder T, De Soyza A, Diar Bakerly N, Easom N, Geddes JR, Greening NJ, Hart N, Heaney LG, Heller S, Howard L, Hurst JR, Jacob J, Jenkins RG, Jolley C, Kerr S, Kon OM, Lewis K, Lord JM, McCann GP, Neubauer S, Openshaw PJM, Parekh D, Pfeffer P, Rahman NM, Raman B, Richardson M, Rowland M, Semple MG, Shah AM, Singh SJ, Sheikh A, Thomas D, Toshner M, Chalmers JD, Ho LP, Horsley A, Marks M, Poinasamy K, Wain LV, Brightling CE; PHOSP-COVID Collaborative Group. Physical, cognitive, and mental health impacts of COVID-19 after hospitalisation (PHOSP-COVID): a UK multicentre, prospective cohort study. Lancet Respir Med. 2021 Nov;9(11):1275-1287. doi: 10.1016/S2213-2600(21)00383-0. Epub 2021 Oct 7. PMID 34627560
- [Background] Iadecola C, Anrather J, Kamel H. Effects of COVID-19 on the Nervous System. Cell. 2020 Oct 1;183(1):16-27.e1. doi: 10.1016/j.cell.2020.08.028. Epub 2020 Aug 19. PMID 32882182
- [Background] Cheuk DK, Yeung WF, Chung KF, Wong V. Acupuncture for insomnia. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD005472. doi: 10.1002/14651858.CD005472.pub3. PMID 22972087
- [Background] Lin CC, Chen MC, Yu SN, Ju MS. Chronic electrical stimulation of four acupuncture points on rat diabetic neuropathy. Conf Proc IEEE Eng Med Biol Soc. 2005;2005:4271-4. doi: 10.1109/IEMBS.2005.1615408. PMID 17281178
- [Background] Ji S, Duan J, Hou X, Zhou L, Qin W, Niu H, Luo S, Zhang Y, Chan P, Jin X. The Role of Acupuncture Improving Cognitive Deficits due to Alzheimer's Disease or Vascular Diseases through Regulating Neuroplasticity. Neural Plast. 2021 Jan 12;2021:8868447. doi: 10.1155/2021/8868447. eCollection 2021. PMID 33505460
- [Background] Pei W, Meng F, Deng Q, Zhang B, Gu Y, Jiao B, Xu H, Tan J, Zhou X, Li Z, He G, Ruan J, Ding Y. Electroacupuncture promotes the survival and synaptic plasticity of hippocampal neurons and improvement of sleep deprivation-induced spatial memory impairment. CNS Neurosci Ther. 2021 Dec;27(12):1472-1482. doi: 10.1111/cns.13722. Epub 2021 Oct 8. PMID 34623740
- [Background] Gong, Y., Si, X., & Zhang, Y. (2021). Clinical application and practice of acupuncture therapy in COVID- 19. Zhongguo Zhen Jiu, 41, 142-4.
- [Background] Liu WH, Guo SN, Wang F, Hao Y. Understanding of guidance for acupuncture and moxibustion interventions on COVID-19 (Second edition) issued by CAAM. World J Acupunct Moxibustion. 2020 Mar;30(1):1-4. doi: 10.1016/j.wjam.2020.03.005. Epub 2020 Mar 17. PMID 32292259
- [Background] Jia H, Han Z, Zhang K, Tang Q, Sun K, Huang H, Qi F. Acupuncture and related interventions for anxiety in coronavirus disease 2019: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Jul 24;99(30):e21317. doi: 10.1097/MD.0000000000021317. PMID 32791723
- [Background] von Trott P, Oei SL, Ramsenthaler C. Acupuncture for Breathlessness in Advanced Diseases: A Systematic Review and Meta-analysis. J Pain Symptom Manage. 2020 Feb;59(2):327-338.e3. doi: 10.1016/j.jpainsymman.2019.09.007. Epub 2019 Sep 18. PMID 31539602
- [Background] Zhang K, Gao C, Li C, Li Y, Wang S, Tang Q, Zhao C, Zhai J. Acupuncture for Acute Pancreatitis: A Systematic Review and Meta-analysis. Pancreas. 2019 Oct;48(9):1136-1147. doi: 10.1097/MPA.0000000000001399. PMID 31593017
- [Background] Han Z, Zhang Y, Wang P, Tang Q, Zhang K. Is acupuncture effective in the treatment of COVID-19 related symptoms? Based on bioinformatics/network topology strategy. Brief Bioinform. 2021 Sep 2;22(5):bbab110. doi: 10.1093/bib/bbab110. PMID 33866350
- [Background] Zhang B, Zhang K, Tang Q, Sun K, Han Z. Acupuncture for breathlessness in COVID-19: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Jul 2;99(27):e20701. doi: 10.1097/MD.0000000000020701. PMID 32629642
- [Background] Zhang Q, Xu X, Sun S, Cao F, Li J, Qi X, Ji G, Wang Y, Song B. Efficacy of acupuncture and moxibustion in adjuvant treatment of patients with novel coronavirus disease 2019 (COVID-19): A protocol for systematic review and meta analysis. Medicine (Baltimore). 2020 Jul 10;99(28):e21039. doi: 10.1097/MD.0000000000021039. PMID 32664113
- [Background] He W, Li M, Han X, Zhang W. Acupuncture for Mild Cognitive Impairment and Dementia: An Overview of Systematic Reviews. Front Aging Neurosci. 2021 May 14;13:647629. doi: 10.3389/fnagi.2021.647629. eCollection 2021. PMID 34054504
- [Background] Su XT, Wang LQ, Li JL, Zhang N, Wang L, Shi GX, Yang JW, Liu CZ. Acupuncture Therapy for Cognitive Impairment: A Delphi Expert Consensus Survey. Front Aging Neurosci. 2020 Nov 26;12:596081. doi: 10.3389/fnagi.2020.596081. eCollection 2020. PMID 33328975
- [Background] White AR, Filshie J, Cummings TM; International Acupuncture Research Forum. Clinical trials of acupuncture: consensus recommendations for optimal treatment, sham controls and blinding. Complement Ther Med. 2001 Dec;9(4):237-45. doi: 10.1054/ctim.2001.0489. PMID 12184353
- [Background] Sun Y, Liu Y, Liu B, Zhou K, Yue Z, Zhang W, Fu W, Yang J, Li N, He L, Zang Z, Su T, Fang J, Ding Y, Qin Z, Song H, Hu H, Zhao H, Mo Q, Zhou J, Wu J, Liu X, Wang W, Pang R, Chen H, Wang X, Liu Z. Efficacy of Acupuncture for Chronic Prostatitis/Chronic Pelvic Pain Syndrome : A Randomized Trial. Ann Intern Med. 2021 Oct;174(10):1357-1366. doi: 10.7326/M21-1814. Epub 2021 Aug 17. PMID 34399062
- [Background] Tu JF, Yang JW, Shi GX, Yu ZS, Li JL, Lin LL, Du YZ, Yu XG, Hu H, Liu ZS, Jia CS, Wang LQ, Zhao JJ, Wang J, Wang T, Wang Y, Wang TQ, Zhang N, Zou X, Wang Y, Shao JK, Liu CZ. Efficacy of Intensive Acupuncture Versus Sham Acupuncture in Knee Osteoarthritis: A Randomized Controlled Trial. Arthritis Rheumatol. 2021 Mar;73(3):448-458. doi: 10.1002/art.41584. Epub 2021 Jan 15. PMID 33174383
- [Background] Tan TT, Wang D, Huang JK, Zhou XM, Yuan X, Liang JP, Yin L, Xie HL, Jia XY, Shi J, Wang F, Yang HB, Chen SJ. Modulatory effects of acupuncture on brain networks in mild cognitive impairment patients. Neural Regen Res. 2017 Feb;12(2):250-258. doi: 10.4103/1673-5374.200808. PMID 28400807
- [Background] Whiting M, Leavey G, Scammell A, Au S, King M. Using acupuncture to treat depression: a feasibility study. Complement Ther Med. 2008 Apr;16(2):87-91. doi: 10.1016/j.ctim.2007.07.005. Epub 2007 Sep 29. PMID 18514910
- [Background] Zheng YP, Lin KM. Comparison of the Chinese Depression Inventory and the Chinese version of the Beck Depression Inventory. Acta Psychiatr Scand. 1991 Dec;84(6):531-6. doi: 10.1111/j.1600-0447.1991.tb03189.x. PMID 1792927
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Fang J, Chen L, Ma R, Keeler CL, Shen L, Bao Y, Xu S. Comprehensive rehabilitation with integrative medicine for subacute stroke: A multicenter randomized controlled trial. Sci Rep. 2016 May 13;6:25850. doi: 10.1038/srep25850. PMID 27174221